CLINICAL TRIAL: NCT00968448
Title: Inspiratory Muscle Training (IMT) in Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Prof. Tim Meyer, Saarland University
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Sportmed-Saarland-8/2009
Record Dates: First submitted 2009-08-28; First posted 2009-08-31 (Estimated); Last update posted 2011-01-05 (Estimated); Status verified 2009-08

CONDITIONS: Running Endurance
Keywords: respiratory muscle; breathing pattern; exercise performance
MeSH Terms: interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Training (Active Comparator): respiratory muscle training (pressure threshold loading)
  Interventions: Behavioral: Respiratory muscle training
- sham training (Sham Comparator): training with low resistance
  Interventions: Behavioral: Sham training

INTERVENTIONS:
Behavioral: Respiratory muscle training — Daily training with a handheld device (Pressure threshold loading). 1x50 breaths with adjustments (gradually increasing levels).
  Arms: Training
Behavioral: Sham training — Sham training with same handheld device. 50 breaths daily on the lowest level
  Arms: sham training

SUMMARY:
The purpose of this study is to determine weather well trained athletes benefit from inspiratory (respiratory) muscle training.

DETAILED DESCRIPTION:
* Subject: The investigators intend to include 40 well trained runners, 18 years or older.
* Design: Following lung function and exercise testing (incremental treadmill test to exhaustion, 5000m run time trial) participants will be randomly assigned to a verum or a control group. The verum group will train with a hand-held, commercially available pressure threshold loading device (POWERbreathe,UK). The control group will perform a sham-training with the same device. After six to eight weeks the the initial tests will be repeated.
* Hypothesis: Inspiratory muscle training enhances performance on submaximal work loads and in the 5000m run time trial by changes in breathing pattern. Maximum oxygen uptake remains unchanged.

ELIGIBILITY:
Inclusion Criteria:

* well trained runners

Exclusion Criteria:

* previous respiratory muscle training
* cardiovascular diseases
* impaired lung function

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
performance in the 500m run time trial | 6-8 weeks

SECONDARY OUTCOMES:
maximum inspiratory pressure | 6-8- weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Such, MD, Principal Investigator — Institute for Sports Medicine and Prevention / Saarland Universitiy
Locations (1):
- Universität des Saarlands, Saarbrücken, Saarland, Germany